CLINICAL TRIAL: NCT01485536
Title: A Phase II Study of the HSP90 Inhibitor AUY922 in Patients With Relapsed and Refractory Lymphoma
Brief Title: A Study of the HSP90 Inhibitor AUY922
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study halted early due to limited response.
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2011-0467; NCI-2012-00070 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2011-11-29; First posted 2011-12-05 (Estimated); Results first posted 2017-01-23 (Estimated); Last update posted 2017-01-23 (Estimated); Status verified 2015-12

CONDITIONS: Lymphoma
Keywords: Lymphoma; Relapsed/refractory lymphoma; AUY922
MeSH Terms: conditions — Lymphoma | interventions — 5-(2,4-dihydroxy-5-isopropylphenyl)-4-(4-morpholin-4-ylmethylphenyl)isoxazole-3-carboxylic acid ethylamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- AUY922 (Experimental): AUY922 starting dose 70 mg/m2 intravenous on Days 1, 8, 15, and 22 of 28 day cycle.
  Interventions: Drug: AUY922

INTERVENTIONS:
Drug: AUY922 — Starting Dose: 70 mg/m2 by vein on days 1, 8, 15, and 22 days of a 28 day cycle.

SUMMARY:
The goal of this clinical research study is to learn if AUY922 can help to control refractory or recurrent lymphoma. The safety of AUY922 will also be studied.

AUY922 is designed to block tumor growth by blocking a protein.

DETAILED DESCRIPTION:
Study Drug Administration:

If you are found to be eligible to take part in this study, you will receive AUY922 by vein over about 1 hour on Days 1, 8, 15, and 22 of each 28-day cycle.

Study Visits:

On Days 1 and 15 of Cycles 1-12:

* You will have a physical exam, including measurement of your vital signs (blood pressure, heart rate, temperature, and breathing rate).
* Your performance status will be recorded.
* You will be asked about any drugs you may be taking and any side effects you may have had.
* Blood (about 6-7 teaspoons) will be drawn for routine tests. On Day 1 of Cycle 1, this blood will also be used to check your heart function.
* You will have ECGs before and after the study drug infusion.

On Day 8 of Cycles 1-12:

* Your vital signs will be measured.
* You will be asked about any drugs you may be taking and any side effects you may have had.
* Blood (about 6-7 teaspoons) will be drawn for routine tests and to check your heart function.
* You will have ECGs before and after the study drug infusion.

On Day 1 of Cycles 1 and 2:

* Urine will be collected for routine tests.
* Blood (about 1 teaspoon) will be drawn to check your blood clotting function.

On Days 2 and 3 of Cycle 1:

* Blood (about 5-6 teaspoons) will be drawn for routine tests.
* You will have ECGs at about 24 and 48 hours after the end of the infusion.
* You will be asked about any drugs you may be taking, any side effects you may be having, and about your overall health.

On Day 22 of Cycle 1:

* You will have a physical exam, including measurement of your vital signs.
* Your performance status will be recorded.
* You will be asked about any drugs you may be taking, any side effects you may be having, and about your overall health.
* Blood (about 5-6 teaspoons) will be drawn for routine tests.

After every 2 cycles:

* You will have CT and PET scans to check the status of the disease.
* You will be asked about any side effects you may be having and about your overall health.

Anytime the study doctor thinks it is needed, you will have an eye exam or other tests.

Length of Study:

You may continue taking AUY922 for up to 12 cycles. You will no longer be able to take the study drug if the disease gets worse, if intolerable side effects occur, or if you are unable to follow study directions.

End-of-Treatment Visit:

At 28 days after your last dose:

* Blood (about 5-6 teaspoons) and urine will be collected for routine tests.
* Blood (about 1 teaspoon) will be drawn to check your blood clotting function.
* You will have a physical exam, including measurement of your vital signs.
* Your performance status will be recorded.
* You will have an eye exam by an eye doctor.
* You will have CT and PET scans to check the status of the disease.
* You will be asked about any drugs you may be taking, any side effects you may be having, and about your overall health.

Long-Term Follow-Up:

After you stop the study drug, you will have a CT scan and physical exam every 3 months for 1 year, then every 4 months for another year, and every 6 months for 3 years and then 1 time a year after that.

This is an investigational study. AUY922 is not FDA approved or commercially available. It is currently being used for research purposes only.

Up to 42 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Age >/= 18 years
2. Able to sign Informed Consent
3. Patients must have the following laboratory values: Hematologic: Absolute Neutrophil Count (ANC) >/=1.5x10^9/L; Hemoglobin (Hgb) >/=9 g/dl; Platelets (plt) >/=50 x10^9/L. Biochemistry: Potassium within normal limits; Total calcium (corrected for serum albumin) and Phosphorus within normal limits o Magnesium above LLN or correctable with supplements; Liver and Kidney Functions: aspartate aminotransferase (AST)/serum glutamate oxaloacetate transaminase (SGOT) and ALT/serum glutamate pyruvate transaminase (SGPT) </=1.5 x Upper Limit of Normal (ULN) if Alkaline Phosphate (AP) > 2.5 ULN AST/SGOT and ALT/SGPT </=2.5 x Upper Limit of Normal (ULN) if Alkaline Phosphate (AP) </=5.0 x ULN if liver metastases are present; Serum bilirubin </= 1.5 x ULN; Serum creatinine </=1.5 x ULN or 24-hour clearance >/= 50 ml/min.
4. Negative serum pregnancy test. The serum pregnancy test must be obtained prior to the first administration of AUY922 (</= 72 hours prior to dosing) in all pre-menopausal women and women <2 years after the onset of menopause
5. Histologically confirmed Diffuse Large B-cell Lymphoma (DLBCL), (primary mediastinal DLBCL, DLBCL-NOS, large B-cell transformation of indolent B-cell lymphoma including follicular lymphoma, small lymphocytic lymphoma and marginal zone lymphoma) or Peripheral T-cell Lymphoma (PTCL), including PTCL not otherwise specified, angioimmunoblastic lymphoma, anaplastic large T-cell lymphoma, hepatosplenic T-cell lymphoma, enteropathy associated T-cell lymphoma; nodal or extranodal NK/T-cell lymphoma, mycosis fungoides with radiographically measurable disease.
6. Relapsed or refractory after standard treatments and with no curative option with conventional therapy.
7. Measurable disease.
8. No known evidence of cerebral or meningeal involvement by lymphoma.
9. Eastern Cooperative Oncology Group (ECOG) performance status 0 to 2.

Exclusion Criteria:

1. Diarrhea > CTCAE (v4.02) grade 1 that cannot be controlled with oral anti-diarrhea medications.
2. Pregnant or lactating women.
3. Fertile women of childbearing potential (WCBP), a female that has not been surgically sterilized or that has not been amenorrheic for at least 24 consecutive months, not using double-barrier methods of contraception (abstinence, oral contraceptives, intrauterine device or barrier method of contraception in conjunction with spermicidal jelly, or surgically sterile). Male patients whose partners are WCBP not using double-barrier methods of contraception.
4. Impaired cardiac function, including any one of the following: History (or family history) of long QT syndrome; Mean QTc >/= 450 msec on baseline ECG; History of clinically manifested ischemic heart disease </= 6 months prior to study start; History of heart failure or left ventricular (LV) dysfunction (LVEF </=45%) by multigated radionuclide angiography (MUGA) or ECHO; Clinically significant ECG abnormalities including 1 or more of the following: left bundle branch block (LBBB), right bundle branch block (RBBB) with left anterior hemiblock (LAHB). ST segment elevation or depression > 1mm, or 2nd (Mobitz II), or 3rd degree AV block.
5. Continuation #4) History or presence of atrial fibrillation, atrial flutter or ventricular arrhythmias including ventricular tachycardia or Torsades de Pointes; Other clinically significant heart disease (e.g. congestive heart failure, uncontrolled hypertension (2 consecutive reading >140/90), history of labile hypertension, or history of poor compliance with an antihypertensive regimen); Clinically significant resting bradycardia (< 50 beats per minute); Patients who are currently receiving treatment with any medication which has a relative risk of prolonging the QTcF interval or inducing Torsades de Pointes and cannot be switched or discontinued to an alternative drug prior to commencing AUY922;
6. Obligate use of a cardiac pacemaker.
7. All lymphomas except for Diffuse Large B-cell Lymphoma (DLBCL) and Peripheral T-cell Lymphoma (PTCL).
8. Chemotherapy or radiation therapy or other investigational agents within 3 weeks prior to entering the study.
9. Previous radioimmunotherapy within 12 weeks.
10. Patient with known HIV infection.
11. Known active viral hepatitis.
12. Any serious active disease or co-morbid condition, which in the opinion of the principle investigator, will interfere with the safety or with compliance with the study.
13. Serious nonmalignant disease (e.g., congestive heart failure, hydronephrosis); active uncontrolled bacterial, viral, or fungal infections; or other conditions which would compromise protocol objectives in the opinion of the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2012-08; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yasuhiro Oki, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: August 28, 2016 to June 17, 2014. All recruitment done at The University of Texas MD Anderson Cancer Center.
Pre-assignment Details: Of 26 participants screened for enrollment, five were not eligible therefore excluded from the study before any treatment assignment.
Period: Overall Study
Arm/Group | AUY922
Started | 21
Completed | 17
Not Completed | 4
Not completed — Withdrawal by Subject | 3
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | AUY922
Number analyzed (Participants) | 21
Age, Continuous [Median (Full Range); unit: years] | 60 [33 to 77]
Gender [Count of Participants; unit: Participants]
  Female | 5
  Male | 16
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 1
  Black | 1
  Hispanic | 13
  White | 15
Region of Enrollment [Number; unit: participants]
  United States | 21
Baseline Lymphoma Diagnosis [Count of Participants; unit: Participants] — Histologically confirmed participant diagnosis at baseline by Relapsed or Refractory Diffuse Large B-Cell Lymphoma (DLBCL) or peripheral T-cell lymphoma (PTCL)
  Participants
    DLBCL | 14
    PTCL | 6
    Unknown | 1

OUTCOME MEASURES:

1. Primary Outcome: Objective Response in Participants With Relapsed or Refractory Diffuse Large B-cell Lymphoma (DLBCL) and Peripheral T-cell Lymphoma (PTCL)
Description: Objective Response defined as Complete (CR) and Partial (PR) Response. Computed tomography (CT) and Positron emission tomography (PET) scans done after every 2 cycles to assess efficacy using Cheson Criteria (2007) which lists CR as disappearance of all evidence of disease, and PR as regression of measurable disease and no new sites.
Time Frame: 56 days
Population: One participant withdrew therefore was not evaluable for the outcome and is excluded from analysis
Measure: Count of Participants; unit: Participants
Arm/Group | AUY922
Number analyzed (Participants) | 20
Participants
  DLBCL (N=14) | 1
  PTCL (N=6) | 1

2. Primary Outcome: Overall Response Rate (ORR)
Description: Percentage of participants with objective response defined as Complete (CR) and Partial (PR) Response. Computed tomography (CT) and Positron emission tomography (PET) scans done after every 2 cycles to assess efficacy using Cheson Criteria (2007) which lists CR as disappearance of all evidence of disease, and PR as regression of measurable disease and no new sites.
Time Frame: Up to 12 cycles or 48 weeks
Population: One participant withdrew therefore was not evaluable for the outcome and is excluded from analysis
Measure: Number; unit: percentage of participants
Arm/Group | AUY922
Number analyzed (Participants) | 20
percentage of participants
  DLBCL (N=14) | 7
  PTCL (N=6) | 17

ADVERSE EVENTS:
Time Frame: Adverse event data were collected through each four week cycle up to 12 cycles (48 weeks).
Arm/Group | AUY922
Serious Adverse Events (participants affected / at risk) | 4/20
Other Adverse Events (participants affected / at risk) | 20/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AUY922 (N=20)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Thrombocytopenia (Vascular disorders) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Vomiting/Diarrhea (Gastrointestinal disorders) | 1 (1) — Combined incidence of Nausea, Vomiting, Diarrhea
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AUY922 (N=20)
Abdominal pain (Gastrointestinal disorders) | 5 (6)
Activated partial thromboplastin time prolonged (Investigations) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1)
Alkaline phosphatase increased (Investigations) | 1 (1)
Allergic reaction (Immune system disorders) | 1 (1)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Anemia (Blood and lymphatic system disorders) | 9 (16)
Anorexia (Metabolism and nutrition disorders) | 2 (3)
Anxiety (Psychiatric disorders) | 3 (3)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Bloating (Gastrointestinal disorders) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (2)
Blurred vision (Eye disorders) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Bruising (Injury, poisoning and procedural complications) | 1 (1)
Buttock pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Cardiac disorders - (Other) (Cardiac disorders) | 1 (1)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Chills (General disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 6 (6)
Cough (Respiratory, thoracic and mediastinal disorders) | 7 (7)
Creatinine increased (Investigations) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 3 (4)
Depression (Psychiatric disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 10 (23)
Dizziness (Nervous system disorders) | 2 (2)
Dry eye (Eye disorders) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Edema limbs (General disorders) | 6 (6)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 2 (2)
Eye disorders - Impaired vision (Eye disorders) | 7 (13)
Eye infection (Infections and infestations) | 1 (1)
Fatigue (General disorders) | 12 (21)
Fever (General disorders) | 3 (6)
Flashing lights (Eye disorders) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (1)
Floaters (Eye disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1)
Gastrointestinal disorders - (Other) (Gastrointestinal disorders) | 1 (2)
General disorders and administration site conditions - (Other) (General disorders) | 6 (8)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 5 (7)
Headache (Nervous system disorders) | 4 (4)
Hemorrhoids (Gastrointestinal disorders) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 2 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Hypermagnesemia (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 (2)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1)
Hypoglycemia (Metabolism and nutrition disorders) | 2 (2)
Hypokalemia (Metabolism and nutrition disorders) | 4 (5)
Hypomagnesemia (Metabolism and nutrition disorders) | 9 (11)
Hyponatremia (Metabolism and nutrition disorders) | 2 (2)
Hypotension (Vascular disorders) | 4 (5)
Infections and infestations - (Other) (Infections and infestations) | 1 (1)
Insomnia (Psychiatric disorders) | 5 (5)
Investigations - Neutropenia (Investigations) | 1 (1)
Lip infection (Infections and infestations) | 1 (1)
Lung infection (Infections and infestations) | 1 (1)
Malaise (General disorders) | 1 (1)
Mucosal infection (Infections and infestations) | 2 (2)
Mucositis oral (Gastrointestinal disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Nausea (General disorders) | 9 (15)
Nervous system disorders - Numbness & tingling feet (Nervous system disorders) | 1 (1)
Neutrophil count decreased (Investigations) | 5 (10)
Night blindness (Eye disorders) | 2 (2)
Oral pain (Gastrointestinal disorders) | 1 (2)
Pain (General disorders) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7 (7)
Penile infection (Infections and infestations) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 5 (7)
Photophobia (Eye disorders) | 1 (1)
Platelet count decreased (Investigations) | 8 (15)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (3)
Psychiatric disorders - (Other) (Psychiatric disorders) | 1 (1)
Purpura (Skin and subcutaneous tissue disorders) | 1 (1)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory, thoracic and mediastinal disorders - Pneumonia (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Scalp pain (Skin and subcutaneous tissue disorders) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 3 (3)
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Skin and subcutaneous tissue disorders - Lesions (Skin and subcutaneous tissue disorders) | 2 (3)
Social circumstances - Cold Sweat (Social circumstances) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Surgical and medical procedures - Dental procedures (Surgical and medical procedures) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Upper respiratory infection (Infections and infestations) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 1 (1)
Urinary tract infection (Renal and urinary disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 6 (9)
Watering eyes (Eye disorders) | 1 (1)
Weight loss (Investigations) | 2 (2)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2 (2)

LIMITATIONS AND CAVEATS:
Although the study surpassed the first futility endpoint for DLBCL cohort, it was terminated early due to limited responses and significant toxicities witnessed in the entire cohort of the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes